CLINICAL TRIAL: NCT06154837
Title: A Two-part Phase 1 Randomized, Double-blind, Placebo-controlled Study to Investigate Safety, Tolerability, Immunogenicity, Pharmacokinetics and Pharmacodynamics of GSK3862995B Following Single Ascending Doses in Healthy Participants and Repeat Doses in Participants With Chronic Obstructive Pulmonary Disease
Brief Title: A Study for GSK3862995B in Healthy Participants and Participants With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 221531; 2023-506880-32 (Other: EudraCT Number)
Record Dates: First submitted 2023-11-26; First posted 2023-12-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK3862995B; Chronic Obstructive Pulmonary Disease; Phase 1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The primary purpose of the study is to evaluate the safety, and tolerability of GSK3862995B following single dose in healthy participants and repeat doses in participants with Chronic obstructive pulmonary disorder (COPD).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Part A Dose Level 1: Single dose of GSK3862995B (Experimental): Healthy participants will receive single dose of GSK3862995B.
  Interventions: Drug: GSK3862995B
- Part A Dose Level 2: Single dose of GSK3862995B (Experimental): Healthy participants will receive single dose of GSK3862995B.
  Interventions: Drug: GSK3862995B
- Part A Dose Level 3: Single dose of GSK3862995B (Experimental): Healthy participants will receive single dose of GSK3862995B.
  Interventions: Drug: GSK3862995B
- Part A Dose Level 4: Single dose of GSK3862995B (Experimental): Healthy participants will receive single dose of GSK3862995B.
  Interventions: Drug: GSK3862995B
- Part A Dose Level 5: Single dose of GSK3862995B (Experimental): Healthy participants will receive single dose of GSK3862995B.
  Interventions: Drug: GSK3862995B
- Part A Dose Level 6: Single dose of GSK3862995B (Experimental): Healthy participants will receive single dose of GSK3862995B.
  Interventions: Drug: GSK3862995B
- Part A: Placebo (Placebo Comparator): Healthy participants will receive single dose of placebo.
  Interventions: Drug: Placebo
- Part B: Repeat dose of GSK3862995B (Experimental): Participants with COPD will receive repeat doses of GSK3862995B.
  Interventions: Drug: GSK3862995B
- Part B: Placebo (Placebo Comparator): Participants with COPD will receive repeat doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3862995B — GSK3862995B will be administered.
  Arms: Part A Dose Level 1: Single dose of GSK3862995B; Part A Dose Level 2: Single dose of GSK3862995B; Part A Dose Level 3: Single dose of GSK3862995B; Part A Dose Level 4: Single dose of GSK3862995B; Part A Dose Level 5: Single dose of GSK3862995B; Part A Dose Level 6: Single dose of GSK3862995B; Part B: Repeat dose of GSK3862995B
Drug: Placebo — Placebo will be administered.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The primary objective of the study is to investigate the safety and tolerability of ascending doses of GSK3862995B following single dose in healthy participants and repeat doses in participants with Chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

Healthy participants (Part A)

* Participant must be 18 to 65 years of age inclusive.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Body weight within the range 50-110 kilogram (kg) (inclusive)
* Body mass index (BMI) within the range 19.5-32 kilogram per square meter (kg/m^2)
* Male and/or female of non-childbearing potential

Participants with Chronic Obstructive Pulmonary Disorder (COPD) (Part B)

* Participant must be 40 to 75 years of age inclusive.
* Body weight within the range 50-110 kg (inclusive)
* BMI within the range 19.5-32 kg/m^2
* Participant has a confirmed diagnosis of COPD for greater than (>)12 months
* Participants must present with a measured post-salbutamol Forced expiratory volume in 1 second/Forced vital capacity (FEV1/FVC) ratio of less than (<) 0.70 at screening to confirm the diagnosis of COPD and a measured post-salbutamol FEV1 greater than or equal to (>=) 40% of predicted normal values.
* Participants must have a well-documented requirement for optimized standard of care background therapy that includes daily inhaled medication.
* A peripheral blood eosinophil count of >=150 cells/microliter (mcL) at screening
* Former cigarette smokers with a history of cigarette smoking of >=10 pack-years at screening current smokers (includes the use of any type of nicotine containing product), or non-smokers are permitted
* Male and/or female of non-childbearing potential.

Exclusion Criteria:

* Participant has a past or current medical condition(s) or disease(s) that is/are not well controlled and, which in the judgement of the Investigator, may affect participant safety or affect study endpoints.
* A history of recurrent infections, or treatment of a chronic infection within 3 months prior to the first dose of study drug, including both serious local infection (for example, cellulitis, abscess) or systemic infection (for example, pneumonia, tuberculosis, hepatitis B, shingles).
* Significant allergies to humanized monoclonal antibodies.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years
* Alanine transaminase (ALT) >1x upper limit of normal (ULN)
* Total bilirubin >1.5xULN (isolated total bilirubin >1.5xULN is acceptable if total bilirubin is fractionated and direct bilirubin less than (<) 35%).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A clinically significant abnormality in 12-lead ECG readings performed at screening
* A clinically significant abnormality in the Holter monitor performed at screening (IV cohorts only).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 36 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persisting disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment is categorized as SAE.
Part B: Number of Participants with AEs and SAEs | Up to 48 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persisting disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment is categorized as SAE.
Part A: Number of Participants with Clinically significant changes in laboratory values | Up to 28 weeks
  Number of Participants with clinically significant changes in laboratory values (haematology, chemistry, and urinalysis) will be assessed.
Part A: Number of Participants with Clinically Significant Change in vital signs | Up to 28 weeks
  Number of participants with clinically significant change in vital signs (tympanic temperature, pulse rate, respiratory rate, and blood pressure) will be assessed.
Part A: Number of Participants with Clinically Significant Change in 12-lead Electrocardiogram (ECG) Parameters | Up to 28 weeks
  Number of participants with clinically significant change in 12-lead ECG parameters will be assessed.
Part B: Number of Participants with Clinically significant changes in laboratory values (haematology, chemistry and urinalysis) | Up to 42 weeks
  Number of Participants with clinically significant changes in laboratory values (haematology, chemistry and urinalysis) will be assessed.
Part B: Number of Participants with Clinically Significant Change in vital signs | Up to 42 weeks
  Number of participants with clinically significant change in vital signs (tympanic temperature, pulse rate, respiratory rate, and blood pressure) up to end of intervention period will be assessed.
Part B: Number of Participants with Clinically Significant Change in 12-lead Electrocardiogram (ECG) Parameters | Up to 42 weeks
  Number of participants with clinically significant change in 12-lead ECG parameters will be assessed.

SECONDARY OUTCOMES:
Part A: Area Under the Concentration-time Curve to the Last Quantifiable Concentration [AUC(0-t)] | Up to 28 weeks
  Blood samples were collected at the indicated time points for pharmacokinetic (PK) analysis. PK parameters were calculated by standard non-compartmental analysis.
Part A: Area Under the Concentration-time Curve to the Infinity (inf) [AUC(0-inf)] | Up to 28 weeks
  Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis.
Part A: Maximum Concentration (Cmax) | Up to 28 weeks
  Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis.
Part B: Area Under the Concentration-time Curve Over the Dosing Interval [AUC(0-tau)] | Up to 42 weeks
  Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis.
Part B: Cmax | Up to 42 weeks
  Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis.
Part A: Number of Participants with Anti-Drug Antibodies (ADA) against GSK3682995B | Up to 28 weeks
  Blood samples were analyzed for the presence of anti-GSK3682995B antibodies by binding ADA assay.
Part B: Number of participants with Incidence of Anti-Drug Antibodies (ADA) against GSK3682995B | Up to 42 weeks
  Blood samples were analyzed for the presence of anti-GSK3682995B antibodies by binding ADA assay.
Part A: Ratio to Baseline in Absolute and Relative Blood Eosinophil Count | Baseline and up to 28 weeks
  Ratio to baseline in absolute and relative blood eosinophil count will be assessed.
Part B: Ratio to Baseline in Absolute and Relative Blood Eosinophil Count | Baseline and up to 42 weeks
  Ratio to baseline in absolute and relative blood eosinophil count will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (9):
  - GSK Investigational Site, Yuma, Arizona
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Austin, Texas
- Germany (12):
  - GSK Investigational Site, Ahrensburg
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Immenhausen
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Lübeck
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, München
  - GSK Investigational Site, Schwerin
- United Kingdom (7):
  - GSK Investigational Site, Barnsley
  - GSK Investigational Site, Blackpool
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Cannock
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/